CLINICAL TRIAL: NCT00641277
Title: A Study to Evaluate the Efficacy of the 3mm Maximus Dental Implant in Areas of Limited Tooth-to-tooth Spacing
Brief Title: Longitudinal Efficacy of Dental Implants in Anterior Areas
Acronym: Maximus
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Reddy, DMD, Dean, School of Dentistry, University of Alabama at Birmingham
Other Study IDs: W040218006
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Edentulous
Keywords: endosseous dental implants; dental aesthetics
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dental implants are used in dentistry to reestablish function and appearance to areas of the mouth where natural teeth are missing. Implants can be a good choice for almost all areas of the mouth except where the space left by missing teeth is too narrow. This is usually the case when front teeth are lost of have been missing since birth.

The Maximus dental implant is the smallest implant made, just 3mm in diameter, and is especially designed to replace missing front teeth and yet be strong enough to function as a natural tooth.

This study will assess the functional success of BioHorizons Maximus one-piece endosseous dental implant.

We hypothesize that placement of the 3mm dental implant in areas of limited tooth-to-tooth spacing will be an efficacious tooth root replacement.

DETAILED DESCRIPTION:
When maxillary anterior (upper front)and/or mandibular incisors are congenitally missing or lost due to other causes, the space between adjacent teeth is frequently too narrow to support traditional implant therapy and patients are often advised to fill the space with conventional fixed or removable prosthetic appliances.

The one-piece titanium construction of the Maximus design is believed to retain optimal biomechanical stength while remaining small enough for use in anterior reconstruction thereby allowing access to spaces that were previously beyond the scope of implant dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Missing anterior teeth

Exclusion Criteria:

* Pregnancy
* Cigarette smoking
* Diabetes Mellitus
* Other significant medical conditions or habits likely to compromise bone healing
* Chronic use of medications likely to compromise bone healing

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2004-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
peri-implant bone support | 5 years following prosthetic attachment

SECONDARY OUTCOMES:
Aesthetics and function | 5 years following prosthectic attachment

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, DMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama, United States

REFERENCES:
- [Background] Branemark PI, Adell R, Breine U, Hansson BO, Lindstrom J, Ohlsson A. Intra-osseous anchorage of dental prostheses. I. Experimental studies. Scand J Plast Reconstr Surg. 1969;3(2):81-100. doi: 10.3109/02844316909036699. No abstract available. PMID 4924041
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] Adell R, Eriksson B, Lekholm U, Branemark PI, Jemt T. Long-term follow-up study of osseointegrated implants in the treatment of totally edentulous jaws. Int J Oral Maxillofac Implants. 1990 Winter;5(4):347-59. PMID 2094653
- [Background] Albrektsson T, Dahl E, Enbom L, Engevall S, Engquist B, Eriksson AR, Feldmann G, Freiberg N, Glantz PO, Kjellman O, et al. Osseointegrated oral implants. A Swedish multicenter study of 8139 consecutively inserted Nobelpharma implants. J Periodontol. 1988 May;59(5):287-96. doi: 10.1902/jop.1988.59.5.287. PMID 3290429
- [Background] Albrektsson T. On long-term maintenance of the osseointegrated response. Aust Prosthodont J. 1993;7 Suppl:15-24. PMID 8054223
- [Background] Engquist B, Bergendal T, Kallus T, Linden U. A retrospective multicenter evaluation of osseointegrated implants supporting overdentures. Int J Oral Maxillofac Implants. 1988 Summer;3(2):129-34. No abstract available. PMID 3075194
- [Background] Jemt T, Lekholm U, Adell R. Osseointegrated implants in the treatment of partially edentulous patients: a preliminary study on 876 consecutively placed fixtures. Int J Oral Maxillofac Implants. 1989 Fall;4(3):211-7. PMID 2700745
- [Background] Buser D, Mericske-Stern R, Bernard JP, Behneke A, Behneke N, Hirt HP, Belser UC, Lang NP. Long-term evaluation of non-submerged ITI implants. Part 1: 8-year life table analysis of a prospective multi-center study with 2359 implants. Clin Oral Implants Res. 1997 Jun;8(3):161-72. doi: 10.1034/j.1600-0501.1997.080302.x. PMID 9586460
- [Background] Wedgwood D, Jennings KJ, Critchlow HA, Watkinson AC, Shepherd JP, Frame JW, Laird WR, Quayle AA. Experience with ITI osseointegrated implants at five centres in the UK. Br J Oral Maxillofac Surg. 1992 Dec;30(6):377-81. doi: 10.1016/0266-4356(92)90204-v. PMID 1450160